CLINICAL TRIAL: NCT04159363
Title: The Effectiveness of an Interactive Colorectal Cancer Self-Management Enhancement Smartphone-based Psychosocial Intervention Programme (iCanManage) on Outcomes of Patients With Colorectal Cancer and Their Family Caregivers
Brief Title: A Psychosocial Intervention for Patients With Colorectal Cancer and Their Family Caregivers
Acronym: iCanManage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore Cancer Society (Other)
Collaborators: National University Hospital, Singapore (Other); Singapore General Hospital (Other)
Responsible Party: Principal Investigator, HE Hong-Gu, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SCS2018
Record Dates: First submitted 2019-10-15; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer
Keywords: psychosocial intervention; smartphone-based; patient; colorectal cancer; caregiver; randomised controlled trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive an interactive Colorectal Cancer self-Management enhancement smartphone-based psychosocial intervention programme (iCanManage) in addition to routine care provided by the respective hospitals.
  Interventions: Other: An interactive Colorectal Cancer self-Management enhancement smartphone-based psychosocial intervention programme (iCanManage)
- Control group (No Intervention): Participants in the control group will receive routine care provided by the respective hospitals . The routine care includes normal consultation with their attending physician, information concerning treatment plans, such as surgical procedures and its associated risks, preoperative preparations and postoperative care, treatment after discharge and/or subsequent adjunct therapy if required.

INTERVENTIONS:
Other: An interactive Colorectal Cancer self-Management enhancement smartphone-based psychosocial intervention programme (iCanManage) — The iCanManage consists of two components: (1a) Existing functions from the BuddyCare mobile application that provide a comprehensive 29 day-by-day perioperative guide for patients who will be undergoing colorectal elective surgery; (1b) a dashboard for healthcare professionals to monitor patients and their caregivers' well-being as well as allow mutual communication; and (2) Newly developed digitalised psychosocial content (e.g., mindfulness-based activities with audio cover, video materials related to positive psychology, patient ambassadors' success stories and relevant psychoeducation) tailored for colorectal cancer patients and caregivers, with the aim of providing them emotional and psychosocial support.
  Arms: Intervention group

SUMMARY:
This study aims to develop a smartphone-based psychosocial intervention for patients with colorectal cancer and their family caregivers and to improve patients' confidence in self-care, psychological well-being, social support, quality of life, and satisfaction with care, as well as caregivers' burden, psychological well-being, and quality of life. The study also aims to explore patients' and their caregivers' perceptions of the intervention and routine care. A multi-centre two-arm experimental study design is used in this study. A total of 100 patient-caregiver dyads will be recruited and randomly allocated to either the control group (receiving routine care alone) or the intervention group (receiving routine care plus the psychosocial intervention). After completed the study, 15 patient-caregiver dyads will be invited for interviews to explore their perceptions on the intervention and/or routine care. This study will generate evidence on the effectiveness of the easily accessible and sustainable smartphone-based psychosocial intervention.

DETAILED DESCRIPTION:
1. Aims The aims of the study are: (1) To develop an interactive Colorectal Cancer self-Management enhancement smartphone-based psychosocial intervention programme (iCanManage program); (2) To examine the effectiveness of iCanManage for colorectal cancer patients and their caregivers in improving patients' health outcomes including self-efficacy (primary outcome), psychological well-being (anxiety & depression), social support, health-related quality of life (HRQoL) and satisfaction with care, as well as caregivers' burden, psychological well-being, and quality of life (QoL) (primary outcome); and (3) To explore patients' and their caregivers' perceptions of iCanManage and routine care.
2. Hypotheses Over 3 months' follow-up, compared to patients in the control group,patients who receive iCanManage in addition to hospital routine care will report significantly: (1) higher levels of self-efficacy, social support, HRQoL and satisfaction with care, and (2) lower levels of anxiety and depression; whilst caregivers will report significantly lower levels of burden, anxiety and depression, and higher level of QoL.
3. Methodology A multi-centre two-arm randomised controlled trial will be conducted at two public hospitals in Singapore. A total of 100 patient-caregiver dyads will be recruited via convenience sampling. Participants (patient-caregiver dyads) will be randomly allocated to either the intervention (receiving iCanManage in addition to hospital routine care) or the control group (receiving only hospital routine care). The aforementioned outcomes of both patients and caregivers will be measured at baseline (start of access to iCanManage), 2-weeks post-surgery (end of access to iCanManage) and 3-months post-surgery. Descriptive statistics, repeated measures analysis of covariance, univariate analysis of covariance (ANCOVA) will be used to analyse the data. At the end of the trial, semi-structured interviews will be conducted to explore 30 patients' and 30 caregivers' perceptions on iCanManage and or routine care. The transcribed interview data will be analysed using a thematic analysis.
4. Significance of the study This study will generate evidence on the effectiveness of the easily accessible and sustainable iCanManage. Should the quantitative and qualitative findings support the feasibility and effects of the intervention, it can be adopted by hospital policymakers as added routine care to enhance patients' self-management ability throughout their surgery journey.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for patients are:

  1. Aged 21 years old and above;
  2. Diagnosed with primary colorectal cancer;
  3. Scheduled for elective colorectal surgeries;
  4. Able to read and speak English and/or Mandarin;
  5. Have a smartphone with internet access; and
  6. Have one identifiable main family caregiver

The inclusion criteria for caregivers include:

1. Aged 21 years old and above;
2. Main family caregiver of the patient
3. Able to read and speak English and/or Mandarin; and
4. Have a smartphone with internet access

Exclusion Criteria for both patients and caregivers:

1. visual or hearing impairments; and/or
2. cognitive impairments/mental disorders identified in their medical record

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer patients' self-efficacy | Patients' self-efficacy will be assessed at baseline (around 2 weeks before surgery) and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  The level of patient's self-efficacy will be measured by the 10-item General Self-Efficacy Scale (GSE). The General Self-Efficacy (GSE) Scale is a 4-point Likert scale (1 = not at all true, 2 = hardly true, 3 = moderately true, 4 = exactly true). The sum score ranges between 10 and 40 with a higher score indicating more self-efficacy.
Caregivers' quality of life | Caregivers' quality of life will be assessed at baseline (around 2 weeks before surgery) and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  Caregivers' quality of life will be measured by 35-item Caregiver Quality of Life Index Cancer (CQOLC). Each item is scored from 0 (not at all) to 4 (very much). The total possible score is 140, with higher scores representing better quality of life.

SECONDARY OUTCOMES:
Patients' anxiety and depression | will be assessed at baseline (around 2 weeks before surgery) and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  Patients' anxiety and depression will be measured by the 14-item Hospital Anxiety and Depression scale (HADS). The Hospital Anxiety and Depression Scale comprises of 14-item self-report scale, 7 items for anxiety and 7 for depression. Each item on the HADS was scored on a four point (0-3) so the possible scores ranged from 0-21 for anxiety and 0-21 for depression. The scores of 8-10 in each scale may be suggestive of borderline risk of anxiety or depression and 11 or higher were indicative of probable 'caseness' of anxiety or depression (Pritchard, 2011; Snaith, 2003).
Patients' Social support | Patients' social support will be assessed at baseline (around 2 weeks before surgery) and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  The level of patients social support will be measured by the 19-item Medical Outcomes Study Social Support Survey (MOS-SSS). The Medical Outcomes Study Social Support Survey (MOS - SSS) measures four aspects of social support including (1) tangible support; (2) affectionate support; (3) positive social interaction and (4) emotional-informational support (Shebourne & Stewart, 1991; Wang, Zheng, He, & Thompson, 2013). Without regarding the source of support, the frequency of support available to each participant was captured through response indications from none-of-the-time (= 1) to all-of-the-time (= 5) on a 5-point scale. Tabulated scores for each dimension are then rescaled to a 0 to 100 range, where higher scores indicate higher support availability (McDowell, 2006).
Patients' Health-related quality of life | Patients' health-related quality of life will be assessed at baseline (around 2 weeks before surgery) and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  Patients' health-related quality of life will be measured by the 29-item European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Colorectal cancer specific (EORTC QLQ-CR29). The EORTC QLQ-CR29 has 29 questions comprises of four functional scales and 18 symptoms scales. All the items are scored on a four-point Likert scale (1-4). Raw scores will be linearly transformed to a scale scores ranging from 0 to100 according to EORTC scoring manual (Fayers et al., 2001). A high scale score for functional scale represents a better functioning, while a high score for a symptom scale represents a worse symptom.
Patients' Satisfaction with care | Patients' satisfaction with care will be assessed at baseline (around 2 weeks before surgery) ,and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  Patients' satisfaction with care will be measured by the 1-item 6-point Ordinal Descriptive Scale (ODS) from 1 (very dissatisfied) to 6 (very satisfied).
Caregivers' burden | Caregivers' burden will be assessed at baseline (around 2 weeks before surgery) and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  Caregivers' burden will be measured by the 21-item Caregiver Reaction Assessment (CRA). The CRA contains subscales of self-esteem, family support, finances, schedule, and health. Each item is scored on a five-point Likert scale, ranging from strongly disagree (score 1) to strongly agree (score 5). The items constituting a particular subscale are averaged to generate subscale scores (ranging from 1 to 5). A higher score on the self-esteem subscale indicates a more positive effect of caregiving, higher scores on the other subscales indicate greater negative effects of caregiving in those domains.
Caregivers' anxiety and depression | Caregivers' anxiety and depression will be assessed at baseline (around 2 weeks before surgery) and assessing changes between baseline and around 2 weeks after the surgery and 3 months after the surgery.
  Caregivers' anxiety and depression will be measured by the 14-item Hospital Anxiety and Depression Scale (HADS). HADS comprises of 14-item self-report scale, 7 items for anxiety and 7 for depression. Each item on the HADS was scored on a four point (0-3) so the possible scores ranged from 0-21 for anxiety and 0-21 for depression. The scores of 8-10 in each scale may be suggestive of borderline risk of anxiety or depression and 11 or higher were indicative of probable 'caseness' of anxiety or depression (Pritchard, 2011; Snaith, 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Gu HE, PhD, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: No
The individual participant data will only be available for researchers involved in this study.

REFERENCES:
- [Background] Al Daken LI, Ahmad MM. The implementation of mindfulness-based interventions and educational interventions to support family caregivers of patients with cancer: A systematic review. Perspect Psychiatr Care. 2018 Jul;54(3):441-452. doi: 10.1111/ppc.12286. Epub 2018 May 10. PMID 29745417
- [Background] Ang SG, Chen HC, Siah RJ, He HG, Klainin-Yobas P. Stressors relating to patient psychological health following stoma surgery: an integrated literature review. Oncol Nurs Forum. 2013 Nov;40(6):587-94. doi: 10.1188/13.ONF.587-594. PMID 24161637
- [Background] Badr H, Lipnick D, Diefenbach MA, Posner M, Kotz T, Miles B, Genden E. Development and usability testing of a web-based self-management intervention for oral cancer survivors and their family caregivers. Eur J Cancer Care (Engl). 2016 Sep;25(5):806-21. doi: 10.1111/ecc.12396. Epub 2015 Oct 27. PMID 26507369
- [Background] Badr H, Carmack CL, Diefenbach MA. Psychosocial interventions for patients and caregivers in the age of new communication technologies: opportunities and challenges in cancer care. J Health Commun. 2015;20(3):328-42. doi: 10.1080/10810730.2014.965369. Epub 2015 Jan 28. PMID 25629218
- [Background] Bandura, A. (1997). Self-efficacy: The Exercise of Control. New York: Freeman.
- [Background] Bazaliński, D., Salacinska, I., Wiech, P. & Kozka, M. (2014). Life satisfaction and self-efficacy in patients with stoma. Progress in Health Sciences, 4(2), 22-30.
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Bevans M, Sternberg EM. Caregiving burden, stress, and health effects among family caregivers of adult cancer patients. JAMA. 2012 Jan 25;307(4):398-403. doi: 10.1001/jama.2012.29. PMID 22274687
- [Background] Butler DL. Early postoperative complications following ostomy surgery: a review. J Wound Ostomy Continence Nurs. 2009 Sep-Oct;36(5):513-9; quiz 520-1. doi: 10.1097/WON.0b013e3181b35eaa. PMID 19752661
- [Background] Raingruber B. The effectiveness of psychosocial interventions with cancer patients: an integrative review of the literature (2006-2011). ISRN Nurs. 2011;2011:638218. doi: 10.5402/2011/638218. Epub 2011 Nov 16. PMID 22191052
- [Background] Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. Health Serv Res. 2007 Aug;42(4):1758-72. doi: 10.1111/j.1475-6773.2006.00684.x. PMID 17286625
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3(2), 77-101.
- [Background] Carlson, L., & Speca, M. (2011). Mindfulness-Based Cancer Recovery: A step-by-step MBSR Approach to help you cope with treatment & reclaim your life. Oakland, CA: New Harbinger Publications.
- [Background] Carter PA. A brief behavioral sleep intervention for family caregivers of persons with cancer. Cancer Nurs. 2006 Mar-Apr;29(2):95-103. doi: 10.1097/00002820-200603000-00003. PMID 16565618
- [Background] Chawla N, Butler EN, Lund J, Warren JL, Harlan LC, Yabroff KR. Patterns of colorectal cancer care in Europe, Australia, and New Zealand. J Natl Cancer Inst Monogr. 2013;2013(46):36-61. doi: 10.1093/jncimonographs/lgt009. PMID 23962509
- [Background] Chenail, R. J. (2011). How to conduct clinical qualitative research on the patient's experience. Qualitative Report, 16(4), 1173-1190.
- [Background] Cotrim H, Pereira G. Impact of colorectal cancer on patient and family: implications for care. Eur J Oncol Nurs. 2008 Jul;12(3):217-26. doi: 10.1016/j.ejon.2007.11.005. PMID 18567538
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Eaton LH, Doorenbos AZ, Schmitz KL, Carpenter KM, McGregor BA. Establishing treatment fidelity in a web-based behavioral intervention study. Nurs Res. 2011 Nov-Dec;60(6):430-5. doi: 10.1097/NNR.0b013e31823386aa. PMID 22048559
- [Background] Fish JA, Ettridge K, Sharplin GR, Hancock B, Knott VE. Mindfulness-based cancer stress management: impact of a mindfulness-based programme on psychological distress and quality of life. Eur J Cancer Care (Engl). 2014 May;23(3):413-21. doi: 10.1111/ecc.12136. Epub 2013 Oct 10. PMID 24118428
- [Background] Fu F, Zhao H, Tong F, Chi I. A Systematic Review of Psychosocial Interventions to Cancer Caregivers. Front Psychol. 2017 May 23;8:834. doi: 10.3389/fpsyg.2017.00834. eCollection 2017. PMID 28596746
- [Background] Gonzalez-Saenz de Tejada M, Bilbao A, Bare M, Briones E, Sarasqueta C, Quintana JM, Escobar A. Association of social support, functional status, and psychological variables with changes in health-related quality of life outcomes in patients with colorectal cancer. Psychooncology. 2016 Aug;25(8):891-7. doi: 10.1002/pon.4022. Epub 2015 Nov 18. PMID 26582649
- [Background] Grassi L, Spiegel D, Riba M. Advancing psychosocial care in cancer patients. F1000Res. 2017 Dec 4;6:2083. doi: 10.12688/f1000research.11902.1. eCollection 2017. PMID 29259774
- [Background] Grimmett C, Haviland J, Winter J, Calman L, Din A, Richardson A, Smith PWF, Foster C. Colorectal cancer patient's self-efficacy for managing illness-related problems in the first 2 years after diagnosis, results from the ColoREctal Well-being (CREW) study. J Cancer Surviv. 2017 Oct;11(5):634-642. doi: 10.1007/s11764-017-0636-x. Epub 2017 Aug 19. PMID 28822053
- [Background] Gustafson DH, DuBenske LL, Namkoong K, Hawkins R, Chih MY, Atwood AK, Johnson R, Bhattacharya A, Carmack CL, Traynor AM, Campbell TC, Buss MK, Govindan R, Schiller JH, Cleary JF. An eHealth system supporting palliative care for patients with non-small cell lung cancer: a randomized trial. Cancer. 2013 May 1;119(9):1744-51. doi: 10.1002/cncr.27939. Epub 2013 Jan 25. PMID 23355273
- [Background] Hildebrandt C, Mayer H, Koller A. Experiences of patients with colorectal cancer from diagnosis until completion of treatment: A meta-ethnography approach. Psychooncology. 2019 Feb;28(2):219-227. doi: 10.1002/pon.4946. Epub 2018 Dec 28. PMID 30447170
- [Background] Huh JW. Stoma Creation After Surgery for Rectal Cancer: Temporary or Permanent? Ann Coloproctol. 2015 Jun;31(3):82. doi: 10.3393/ac.2015.31.3.82. No abstract available. PMID 26161373
- [Background] House JS, Landis KR, Umberson D. Social relationships and health. Science. 1988 Jul 29;241(4865):540-5. doi: 10.1126/science.3399889.
- [Background] Johns SA, Brown LF, Beck-Coon K, Talib TL, Monahan PO, Giesler RB, Tong Y, Wilhelm L, Carpenter JS, Von Ah D, Wagner CD, de Groot M, Schmidt K, Monceski D, Danh M, Alyea JM, Miller KD, Kroenke K. Randomized controlled pilot trial of mindfulness-based stress reduction compared to psychoeducational support for persistently fatigued breast and colorectal cancer survivors. Support Care Cancer. 2016 Oct;24(10):4085-96. doi: 10.1007/s00520-016-3220-4. Epub 2016 May 17. PMID 27189614
- [Background] Kabat-Zinn, J. (2003), Mindfulness-Based Interventions in Context: Past, Present, and Future. Clinical Psychology: Science and Practice, 10: 144-156. doi:10.1093/clipsy.bpg016
- [Background] Kaltenbaugh DJ, Klem ML, Hu L, Turi E, Haines AJ, Hagerty Lingler J. Using Web-based interventions to support caregivers of patients with cancer: a systematic review. Oncol Nurs Forum. 2015 Mar;42(2):156-64. doi: 10.1188/15.ONF.156-164. PMID 25806882
- [Background] Karimi M, Brazier J. Health, Health-Related Quality of Life, and Quality of Life: What is the Difference? Pharmacoeconomics. 2016 Jul;34(7):645-9. doi: 10.1007/s40273-016-0389-9. PMID 26892973
- [Background] Kaynar, G. O. & Vural, F. (2018). Assessment of the caregiver burden of caregivers of colorectal cancer patients. Turkish Journal of Colorectal Disease, 28, 164-171. DOI: 10.4274/tjcd.26121
- [Background] LeSeure P, Chongkham-Ang S. The Experience of Caregivers Living with Cancer Patients: A Systematic Review and Meta-Synthesis. J Pers Med. 2015 Nov 19;5(4):406-39. doi: 10.3390/jpm5040406. PMID 26610573
- [Background] Liao, C. & Qin, Y. (2014). Factors associated with stoma quality of life among stoma patients. International Journal of Nursing Sciences, 1(2), 196 - 201. https://doi.org/10.1016/j.ijnss.2014.05.007
- [Background] Lim, S. H. (2017). Developing and testing the preliminary effects of stoma psychosocial intervention programme on outcomes of colorectal cancer patients with stoma: a mixed methods study. PhD thesis. Singapore: National University of Singapore.
- [Background] Hoon LS, Chi Sally CW, Hong-Gu H. Effect of psychosocial interventions on outcomes of patients with colorectal cancer: a review of the literature. Eur J Oncol Nurs. 2013 Dec;17(6):883-91. doi: 10.1016/j.ejon.2013.05.001. Epub 2013 Jun 4. PMID 23759360
- [Background] Lim SH, Chan SW, He HG. Patients' Experiences of Performing Self-care of Stomas in the Initial Postoperative Period. Cancer Nurs. 2015 May-Jun;38(3):185-93. doi: 10.1097/NCC.0000000000000158. PMID 24836957
- [Background] Loi, T. T. C. (2016). Developing and testing the effects of a psychoeducation intervention on patients with colorectal cancer: a mixed method study. PhD thesis, Singapore: National University of Singapore.
- [Background] Lu LC, Huang XY, Chen CC. The lived experiences of patients with post-operative rectal cancer who suffer from altered bowel function: A phenomenological study. Eur J Oncol Nurs. 2017 Dec;31:69-76. doi: 10.1016/j.ejon.2017.10.004. Epub 2017 Nov 6. PMID 29173830
- [Background] Machin, D., Campbell, M., Fayers, P., & Pinol, A. (1997). Sample size tables for clinical studies (2nd ed.). Oxford: Blackwell Science.
- [Background] Mariotto AB, Yabroff KR, Shao Y, Feuer EJ, Brown ML. Projections of the cost of cancer care in the United States: 2010-2020. J Natl Cancer Inst. 2011 Jan 19;103(2):117-28. doi: 10.1093/jnci/djq495. Epub 2011 Jan 12. PMID 21228314
- [Background] Mehta R, Sharma K, Potters L, Wernicke AG, Parashar B. Evidence for the Role of Mindfulness in Cancer: Benefits and Techniques. Cureus. 2019 May 9;11(5):e4629. doi: 10.7759/cureus.4629. PMID 31312555
- [Background] Melnyk M, Casey RG, Black P, Koupparis AJ. Enhanced recovery after surgery (ERAS) protocols: Time to change practice? Can Urol Assoc J. 2011 Oct;5(5):342-8. doi: 10.5489/cuaj.11002. PMID 22031616
- [Background] Mizuno M, Kakuta M, Ono Y, Kato A, Inoue Y. Experiences of Japanese patients with colorectal cancer during the first six months after surgery. Oncol Nurs Forum. 2007 Jul;34(4):869-76. doi: 10.1188/07.ONF.869-876. PMID 17723988
- [Background] Mosher CE, Adams RN, Helft PR, O'Neil BH, Shahda S, Rattray NA, Champion VL. Family caregiving challenges in advanced colorectal cancer: patient and caregiver perspectives. Support Care Cancer. 2016 May;24(5):2017-2024. doi: 10.1007/s00520-015-2995-z. Epub 2015 Nov 4. PMID 26530227
- [Background] Ni X, Jia D, Chen Y, Wang L, Suo J. Is the Enhanced Recovery After Surgery (ERAS) Program Effective and Safe in Laparoscopic Colorectal Cancer Surgery? A Meta-Analysis of Randomized Controlled Trials. J Gastrointest Surg. 2019 Jul;23(7):1502-1512. doi: 10.1007/s11605-019-04170-8. Epub 2019 Mar 11. PMID 30859422
- [Background] Nikoletti S, Young J, Levitt M, King M, Chidlow C, Hollingsworth S. Bowel problems, self-care practices, and information needs of colorectal cancer survivors at 6 to 24 months after sphincter-saving surgery. Cancer Nurs. 2008 Sep-Oct;31(5):389-98. doi: 10.1097/01.NCC.0000305759.04357.1b. PMID 18772664
- [Background] Northouse L, Kershaw T, Mood D, Schafenacker A. Effects of a family intervention on the quality of life of women with recurrent breast cancer and their family caregivers. Psychooncology. 2005 Jun;14(6):478-91. doi: 10.1002/pon.871. PMID 15599947
- [Background] Northouse LL, Mood DW, Schafenacker A, Montie JE, Sandler HM, Forman JD, Hussain M, Pienta KJ, Smith DC, Kershaw T. Randomized clinical trial of a family intervention for prostate cancer patients and their spouses. Cancer. 2007 Dec 15;110(12):2809-18. doi: 10.1002/cncr.23114. PMID 17999405
- [Background] Ohlsson-Nevo E, Andershed B, Nilsson UG, Anderzen-Carlsson A. Finding a wider horizon: experiences of being a next-of-kin of a person suffering from colorectal cancer as told after having participated in a psychoeducational program. Eur J Oncol Nurs. 2013 Jun;17(3):324-30. doi: 10.1016/j.ejon.2012.09.001. Epub 2012 Oct 1. PMID 23036312
- [Background] Ohlsson-Nevo E, Karlsson J, Nilsson U. Effects of a psycho-educational programme on health-related quality of life in patients treated for colorectal and anal cancer: A feasibility trial. Eur J Oncol Nurs. 2016 Apr;21:181-8. doi: 10.1016/j.ejon.2015.10.002. Epub 2015 Nov 28. PMID 26643400
- [Background] Palma E, Simonetti V, Franchelli P, Pavone D, Cicolini G. An observational study of family caregivers' quality of life caring for patients with a stoma. Gastroenterol Nurs. 2012 Mar-Apr;35(2):99-104. doi: 10.1097/SGA.0b013e31824c2326. PMID 22472669
- [Background] Qian H, Yuan C. Factors associated with self-care self-efficacy among gastric and colorectal cancer patients. Cancer Nurs. 2012 May-Jun;35(3):E22-31. doi: 10.1097/NCC.0b013e31822d7537. PMID 22067688
- [Background] Quinten C, Coens C, Mauer M, Comte S, Sprangers MA, Cleeland C, Osoba D, Bjordal K, Bottomley A; EORTC Clinical Groups. Baseline quality of life as a prognostic indicator of survival: a meta-analysis of individual patient data from EORTC clinical trials. Lancet Oncol. 2009 Sep;10(9):865-71. doi: 10.1016/S1470-2045(09)70200-1. Epub 2009 Aug 18. PMID 19695956
- [Background] Rehse B, Pukrop R. Effects of psychosocial interventions on quality of life in adult cancer patients: meta analysis of 37 published controlled outcome studies. Patient Educ Couns. 2003 Jun;50(2):179-86. doi: 10.1016/s0738-3991(02)00149-0. PMID 12781933
- [Background] Sandelowski M. What's in a name? Qualitative description revisited. Res Nurs Health. 2010 Feb;33(1):77-84. doi: 10.1002/nur.20362. PMID 20014004
- [Background] Schellekens MPJ, van den Hurk DGM, Prins JB, Donders ART, Molema J, Dekhuijzen R, van der Drift MA, Speckens AEM. Mindfulness-based stress reduction added to care as usual for lung cancer patients and/or their partners: A multicentre randomized controlled trial. Psychooncology. 2017 Dec;26(12):2118-2126. doi: 10.1002/pon.4430. Epub 2017 Apr 26. PMID 28337821
- [Background] Schulz KF, Grimes DA. Allocation concealment in randomised trials: defending against deciphering. Lancet. 2002 Feb 16;359(9306):614-8. doi: 10.1016/S0140-6736(02)07750-4. PMID 11867132
- [Background] Shahi V, Lapid MI, Kung S, Atherton PJ, Sloan JA, Clark MM, Rummans TA. Do age and quality of life of patients with cancer influence quality of life of the caregiver? J Geriatr Oncol. 2014 Jul;5(3):331-6. doi: 10.1016/j.jgo.2014.03.003. Epub 2014 Apr 14. PMID 24726867
- [Background] Simmons KL, Smith JA, Bobb KA, Liles LL. Adjustment to colostomy: stoma acceptance, stoma care self-efficacy and interpersonal relationships. J Adv Nurs. 2007 Dec;60(6):627-35. doi: 10.1111/j.1365-2648.2007.04446.x. PMID 18039249
- [Background] Smith F, Ohlen J, Persson LO, Carlsson E. Daily Assessment of Stressful events and Coping in early post-operative recovery after colorectal cancer surgery. Eur J Cancer Care (Engl). 2018 Mar;27(2):e12829. doi: 10.1111/ecc.12829. Epub 2018 Jan 24. PMID 29363821
- [Background] Tamagawa R, Garland S, Vaska M, Carlson LE. Who benefits from psychosocial interventions in oncology? A systematic review of psychological moderators of treatment outcome. J Behav Med. 2012 Dec;35(6):658-73. doi: 10.1007/s10865-012-9398-0. Epub 2012 Jan 22. PMID 22271329
- [Background] Thiele RH, Rea KM, Turrentine FE, Friel CM, Hassinger TE, McMurry TL, Goudreau BJ, Umapathi BA, Kron IL, Sawyer RG, Hedrick TL. Standardization of care: impact of an enhanced recovery protocol on length of stay, complications, and direct costs after colorectal surgery. J Am Coll Surg. 2015 Apr;220(4):430-43. doi: 10.1016/j.jamcollsurg.2014.12.042. Epub 2015 Jan 9. PMID 25797725
- [Background] Thumboo J, Fong KY, Machin D, Chan SP, Soh CH, Leong KH, Feng PH, Thio St, Boey ML. Quality of life in an urban Asian population: the impact of ethnicity and socio-economic status. Soc Sci Med. 2003 Apr;56(8):1761-72. doi: 10.1016/s0277-9536(02)00171-5. PMID 12639592
- [Background] Treanor CJ, Santin O, Prue G, Coleman H, Cardwell CR, O'Halloran P, Donnelly M. Psychosocial interventions for informal caregivers of people living with cancer. Cochrane Database Syst Rev. 2019 Jun 17;6(6):CD009912. doi: 10.1002/14651858.CD009912.pub2. PMID 31204791
- [Background] Waldron EA, Janke EA, Bechtel CF, Ramirez M, Cohen A. A systematic review of psychosocial interventions to improve cancer caregiver quality of life. Psychooncology. 2013 Jun;22(6):1200-7. doi: 10.1002/pon.3118. Epub 2012 Jun 25. PMID 22729992
- [Background] Wang W, Zheng X, He HG, Thompson DR. Psychometric testing of the Chinese Mandarin version of the Medical Outcomes Study Social Support Survey in patients with coronary heart disease in mainland China. Qual Life Res. 2013 Oct;22(8):1965-71. doi: 10.1007/s11136-012-0345-x. Epub 2013 Jan 19. PMID 23334944
- [Background] Wilson IB, Cleary PD. Linking clinical variables with health-related quality of life. A conceptual model of patient outcomes. JAMA. 1995 Jan 4;273(1):59-65. PMID 7996652
- [Background] Worster B, Holmes S. A phenomenological study of the postoperative experiences of patients undergoing surgery for colorectal cancer. Eur J Oncol Nurs. 2009 Dec;13(5):315-22. doi: 10.1016/j.ejon.2009.04.008. Epub 2009 May 30. PMID 19482512
- [Background] Wu HK, Chau JP, Twinn S. Self-efficacy and quality of life among stoma patients in Hong Kong. Cancer Nurs. 2007 May-Jun;30(3):186-93. doi: 10.1097/01.NCC.0000270704.34296.86. PMID 17510581
- [Background] Yabroff KR, Kim Y. Time costs associated with informal caregiving for cancer survivors. Cancer. 2009 Sep 15;115(18 Suppl):4362-73. doi: 10.1002/cncr.24588. PMID 19731345
- [Background] Zhuang CL, Ye XZ, Zhang XD, Chen BC, Yu Z. Enhanced recovery after surgery programs versus traditional care for colorectal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2013 May;56(5):667-78. doi: 10.1097/DCR.0b013e3182812842. PMID 23575408
- [Derived] Wan SW, Chong CS, Toh EL, Lim SH, Loi CT, Lew YFH, Chua MCH, Jee XP, Liu G, Zhu L, Pikkarainen M, He HG. A Theory-Based, Multidisciplinary Approach to Cocreate a Patient-Centric Digital Solution to Enhance Perioperative Health Outcomes Among Colorectal Cancer Patients and Their Family Caregivers: Development and Evaluation Study. J Med Internet Res. 2021 Dec 7;23(12):e31917. doi: 10.2196/31917. PMID 34878991
- See also: Enhanced Recovery after Surgery — https://www.aana.com/practice/clinical-practice-resources/enhanced-recovery-after-surgery
- See also: Singapore Cancer Registry. Cancer Incidence and Mortality 2003 - 2012 and Selected Trends 1973-2012 In Singapore — https://www.nrdo.gov.sg/docs/librariesprovider3/default-document-library/cancertrends_7312_web128e09a5c9d76bafab5aff000014cdee.pdf?sfvrsn=0
- See also: World Health Organization (WHO). Cancer control: diagnosis and treatment. — https://www.who.int/publications-detail/cancer-control-diagnosis-and-treatment